CLINICAL TRIAL: NCT03671187
Title: Effectiveness of Pulmonary Rehabilitation in Smoker Patients With COPD
Brief Title: Pulmonary Rehabilitation and Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof., Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKCU
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Smoking; Rehabilitation; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking (Experimental): 8 week exercise program consists of breathing exercises, strength training and endurance training
  Interventions: Other: Exercise
- Ex- Smoking (Experimental): 8 week exercise program consists of breathing exercises, strength training and endurance training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 8 week exercise program

SUMMARY:
Pulmonary rehabilitation (PR) is known to reduce dyspnea, increase exercise capacity, reduce psychological symptoms and improve quality of life in COPD patients. Some patients continue to smoke despite their illness. Smoking does not create a contraindication to PR. There is insufficient evidence on the effectiveness of PR programs in smoking COPD patients. The purpose of this study, PR completed the program to determine the effectiveness of PR smoker COPD patients.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) is known to reduce dyspnea, increase exercise capacity, reduce psychological symptoms and improve quality of life in COPD patients. Some patients continue to smoke despite their illness. Smoking does not create a contraindication to PR. There is insufficient evidence on the effectiveness of PR programs in smoking COPD patients. The purpose of this study, PR completed the program to determine the effectiveness of PR smoker COPD patients. People who have completed the PR program, smoking and not smoking will be included into the study.

Data of carbon monoxide diffusion test, body plethysmography, 6-min walk test, blood gas analysis, mMRC dyspnea scale, hospital anxiety depression scale, SGRQ and SF-36 quality of life questionnaire performed before and after the program will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients completed 8 PR program

Exclusion Criteria:

* Never smoked patients
* Participated PR program in last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | 6 minutes
  It was performed in a 30-meter long corridor in accordance with American Thoracic

SECONDARY OUTCOMES:
Pulmonary Function Test | 20 minutes
  It was used for assessment of lung functions
Dyspnea Severity | 5 minues
  MMRC Dyspnea Scale (0: no dyspnea, 4: very severe dyspnea), It was used for dyspnea that patients felt during their daily activities.
St. George Disease Related Quality of Life Scale | 20 minutes
  A disease-specific quality of life scale (Max. score:100, lower score means better quality of life level)
Short Form-36 Quality of Life Survey | 25 minutes
  A health related quality of life scale, Short Form-36 Quality of Life Survey (Max. score:100, higher score means better quality of life level)
Hospital Anxiety and Depression Inventory | 20 minutes
  It was used for assessment of anxiety and depression

IPD SHARING:
Plan to Share IPD: No